CLINICAL TRIAL: NCT01737606
Title: Ultrasonic Explorations of Cerebral Tissue Motions - Influence of Aging
Acronym: COSTUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PHAO 2012 - FP / COSTUM
Record Dates: First submitted 2012-11-19; First posted 2012-11-29 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Aging; Cerebral Pulsatility
Keywords: Cerebral pulsatility; Fast Cerebral Pulsatility Imaging or FCPI; MRI; Arteriel Spin Labelling; Cognitive tasks; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- echography (Experimental): Fast Cerebral Pulsatility Imaging
  Interventions: Device: Fast Cerebral Pulsatility Imaging

INTERVENTIONS:
Device: Fast Cerebral Pulsatility Imaging — Cerebral ultrasonic exploration using with neuro-navigation system : 4 acquisitions on 12 or 6 section planes
  Other Names: FCPI

SUMMARY:
The new technical of ultrasonic exploration of this project purpose to validate the measurement of cerebral pulsatility by a new way called "Fast Cerebral Pulsatility Imaging" (FCPI).This will somehow determine the natural history of cerebral pulsatility during development adult to old age

DETAILED DESCRIPTION:
Main objective

Phase 1:

-Study the in-vivo development of ultrasonic method in terms of quality of the acquisitions and intra-operator reproducibility.

Study the ease of positioning in relation to MRI and fusion of MRI and FCPI data via the neuro-navigation system

Phase 2:

-Study the variability of cerebral pulsatility of measured by "Fast Cerebral Pulsatility Imaging" or FCPI with age.

Secondary objectives

* Compare the results of displacements cartography's and vascular cartography obtained by MRI (especially by Arteriel Spin Labelling = ASL)
* Compare results of FCPI with results of cognitive tests of aging separating fluid functions (prefrontal) and functions called crystallized; and study the residual effect of age on cognitive tasks and speed of cognitive processing after taking into account the effect of the cerebral pulsatility
* Compare results of FCPI with electrophysiological measures (PE EEG) describing the attentional control
* Perform an exploratory analysis to highlight the propagating part of the brain displacement maps

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Informed consent form signed
* Person affiliated to a medical insurance
* Male or female
* No smoking the day of the inclusion
* Right handed: Edinburgh test ≥0.8 (subjects of phase 2)
* MMS score ≥ 27 and 5 words score = 10 (subjects of phase 2)
* Socio-educational level greater than or equal to 8 years of school (subjects of phase 2)

Exclusion Criteria:

* Pregnant women, lactating women or women without reliable contraception
* Contraindications to IRM for patients with: ocular metallic foreign object; any electronic medical device implanted by irremovable way (pacemakers, neuro-stimulator, cochlear implants ...); metallic heart valve, old heart valves are specially an absolute contraindication because of risk of dysfunction; vascular clips implanted formerly on brain aneurysm
* Acute medico-surgical condition dating from less than 3 months
* Neurological and neuro-surgical pathology such as: toxic, infectious or inflammatory encephalopathy, epilepsy, intracranial arteriovenous malformation known, intracranial tumor or hydrocephalus known, operated or no, history of ischemic or hemorrhagic stroke, transient or not
* Treatments or pathology that could influence the results of the research: heart failure (dyspnea with stage III or IV NYHA) or non-sinus cardiac rhythm, use of central analgesics or psychotropic drugs
* Psychiatrics disorders of axe 1 of DSM IV, based on MINI (subjects of phase 2)
* Major subject with a legal protection measure
* Subject to exclusion period of any other biomedical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Phase 1 : to validate the technical procedure, we will appreciate several parameters | up to 8 days after consent
  * Time of implementation of procedure
  * Qualitative identification of anatomical landmarks of positioning in space of the US probe using neuro-navigation system; if available quantitative measure: x,y,z or distance to a region of interest(ROI)
  * Perfusion values: Cerebral Blood Flow of Willis' Circle in MRI
  * Signal to noise ratio
  * Amplitude (max displacement value), location (x,y,z of location of this max or distance to a ROI) of FCPI
  * Bandwidth of metrology of FCPI
  * Possibility to indentify the propagation phenomenon underlying to displacements (speed and attenuation of the shear wave)
Phase 2 : the primary outcome measures will be the maximum amplitude and the average amplitude of cerebral movements | up to 8 days after consent
  We hypothesize that the variables describing the FCPI will decrease with age. The primary outcome measures will be the maximum amplitude and the average amplitude of cerebral movements measured in µm in planes chosen previously (for example plan of Circle of Willis and a plane including the dorsolateral area of prefrontal cortex).

SECONDARY OUTCOMES:
Phase 2 : Maps of cerebral displacementand tissular perfusion maps | up to 8 days after consent
  Maps of cerebral displacement obtained by ultrasounds (amplitudes in µm and location in mm) and tissular perfusion maps obtained by Arterial Spin Labelling (Cerebral Blood Flow in µL.g-1.mn-1)
Phase 2 : Measures of FCPI on the regions of interest and cognitive tests | up to 8 days after consent
  Measures of FCPI on the regions of interest: amplitude (maximum displacement values, µm) and location x, y, z, of the location of this maximum in mm, or distance to a region of interest) on the hand and cognitive tests on the other hand expressed with a numerical score for each test.
Phase 2 : Measures of FCPI on the regions of interestand measures of PE EEG | up to 8 days after consent
  Measures of FCPI on the regions of interest: amplitude (maximum displacement values, µm) and location x, y, z, of the location of this maximum in mm, or distance to a region of interest) on the hand and measures of PE EEG on the other hand expressed in terms of amplitude (µV), latency (ms), duration (ms)
Phase 2 : The signal to noise ratio | up to 8 days after consent
  The signal to noise ratio of maps speed (m/s) and attenuation α (cm-1) of the shear wave obtained by mathematical processing of displacement maps

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric PATAT, MD, Principal Investigator — University Hospital of Tours
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Result] Angel L, Bouazzaoui B, Isingrini M, Fay S, Taconnat L, Vanneste S, Ledoux M, Gissot V, Hommet C, Andersson F, Barantin L, Cottier JP, Pasco J, Desmidt T, Patat F, Camus V, Remenieras JP. Brain tissue pulsatility mediates cognitive and electrophysiological changes in normal aging: Evidence from ultrasound tissue pulsatility imaging (TPI). Brain Cogn. 2018 Jun;123:74-80. doi: 10.1016/j.bandc.2018.02.001. Epub 2018 Mar 13. PMID 29544170